CLINICAL TRIAL: NCT05731427
Title: Research on the Mechanism Affecting Progression of Bronchiectasis Based on Omics Method
Brief Title: Research on the Mechanism Affecting Progression of Bronchiectasis
Status: Recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wang xiaorong, Attending physician, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: 2020XHHX002
Record Dates: First submitted 2021-09-15; First posted 2023-02-16 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis; Microbiota; Pseudomonas aeruginosa
MeSH Terms: conditions — Bronchiectasis; Pseudomonas Infections | interventions — Macrolides

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pseudomonas aeruginosa colonization group: Colonization of Pseudomonas aeruginosa in the airways of patients with bronchiectasis
  Interventions: Diagnostic Test: Pseudomonas aeruginosa colonization infection
- Non-Pseudomonas aeruginosa colonization group: No colonization of Pseudomonas aeruginosa in the airways of patients with bronchiectasis
  Interventions: Diagnostic Test: Pseudomonas aeruginosa colonization infection
- Before treatment with macrolides: Before treatment with macrolides in patients with bronchiectasis
  Interventions: Drug: Macrolides
- After treatment with macrolides: After 6 months of treatment with macrolides for patients with bronchiectasis
  Interventions: Drug: Macrolides

INTERVENTIONS:
Diagnostic Test: Pseudomonas aeruginosa colonization infection — With or without airway Pseudomonas aeruginosa colonization infection
  Groups: Non-Pseudomonas aeruginosa colonization group; Pseudomonas aeruginosa colonization group
Drug: Macrolides — Before or after 6 months of treatment with macrolides for patients with bronchiectasis
  Groups: After treatment with macrolides; Before treatment with macrolides

SUMMARY:
Bronchiectasis is a chronic inflammatory respiratory disease defined as the irreversible dilatation of one or more bronchi and is associated with chronic and frequently purulent expectoration, multiple exacerbations and progressive dyspnea. Bronchiectasis has a large heterogeneity. Different patients with bronchiectasis may have different etiology, clinical manifestations, and imaging features. Previous studies showed that there are significant relationship between the airway microbiome and the severity of the disease. For example, patient with airway Pseudomonas aeruginosa colonization has heavier symptoms, heavier severity, poorer quality of life, more acute exacerbations, and worse prognosis. A large number of studies have reported that long-term treatment of low-dose macrolides such as azithromycin or clarithromycin has anti-inflammatory and immunomodulatory effects, which can improve the clinical symptoms and disease progression of various chronic airway diseases, such as diffuse panbronchiolitis, chronic obstructive pulmonary disease, bronchiectasis. Both the 2017 European Respiratory Society guidelines and the 2019 British Thoracic Society Guideline recommend macrolide drugs for the treatment of chronic Pseudomonas aeruginosa colonization bronchiectasis or frequent acute exacerbations bronchiectasis, but the specific mechanism is unknown.This study is based on omics methods (Microbiology and Metabolomics) to deeply explore the composition of airway and gut microbiota in patients with bronchiectasis, the factors affecting the colonization of Pseudomonas aeruginosa and the mechanism of macrolides in the treatment of bronchiectasis.

This project is a multicenter clinical study involving patients with bronchiectasis from Wuhan Union Hospital, Guizhou Provincial People's Hospital, and Yichang Central People's Hospital. Patients with bronchiectasis were recruited according to the inclusion and exclusion criteria. Clinical data were collected from these patients (including demographic information, clinical characteristics, pulmonary function, and lung imaging), along with spontaneously expectorated sputum, feces, and peripheral blood, and the patients were followed for 24 months. The microbiome, metabolome, and cytokines in sputum and feces were assessed, as well as cytokines, inflammatory mediators, and metabolites in peripheral blood.

Through the above methods,investigators further understand the mechanism affecting progression of bronchiectasis and some factors that lead to the colonization of Pseudomonas aeruginosa, as well as mechanisms of macrolides in the treatment of bronchiectasis.

DETAILED DESCRIPTION:
Clinical information:

Demographic information,blood test results,lung function,severity of disease was evaluated using the E-FACED and the Bronchiectasis Severity Index (BSI).The severity of dyspnea was assessed using the Medical Research Council (MRC) grade, and lung radiological severity was assessed using the modified Reiff score and Bhalla score.

Sputum collection:

We collect sputum samples from patients with bronchiectasis. We divided into two parts from each sputum sample, one part was immediately stored -80℃ for microbiota sequencing. The other part was diluted with PBS and centrifuged at 12000g for 5 minutes, and the supernatant was stored at -80°C for measurement of inflammatory factors, oxidative stress and other markers.

Stool collection:

We collect stool samples from patients with bronchiectasis.Fresh stools were processed in the laboratory within 30 min after collection and stored at -80°C until analysis.

Peripheral blood collection:

We collect peripheral blood samples from patients with bronchiectasis to detect inflammatory mediators and so on.

ELIGIBILITY:
Inclusion criteria:

* 18 years or older
* Bronchiectasis confirmed by high-resolution computed tomographic scan(HRCT)
* Chronic expectoration with ability to provide a sputum sample at the study visit
* Provision of written informed consent

Exclusion criteria:

* Traction bronchiectasis
* Lack of important clinical information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with bronchiectasis was recruited from Wuhan Union Hospital.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute exacerbations and mortality | February 10, 2026
  The number of acute exacerbations and outcome (death or survival) of patients with bronchiectasis after one year.

SECONDARY OUTCOMES:
Lung function | February 10, 2026
  Forced expiratory volume in 1s (FEV1),Forced vital capacity（FVC）
Symptoms assessment | February 10, 2026
  MRC score,cough score,sputum purulent score,sputum volume score and hemoptysis score
Stool and sputum microtioba | February 10, 2026
  Stool and sputum microtioba from patients with bronchiectasis after one year

CONTACTS AND LOCATIONS:
Overall Officials: Xiaorong Wang, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (3):
- China (3):
  - Guizhou Provincial people's Hospital, Guiyang, Guizhou
  - Wuhan Union Hospital, Wuhan, Hubei
  - Department of Respiratory and Critical Care Medicine, Yichang Central People's Hospital, Yichang, Hubei

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] De Soyza A, Aksamit T, Bandel TJ, Criollo M, Elborn JS, Operschall E, Polverino E, Roth K, Winthrop KL, Wilson R. RESPIRE 1: a phase III placebo-controlled randomised trial of ciprofloxacin dry powder for inhalation in non-cystic fibrosis bronchiectasis. Eur Respir J. 2018 Jan 25;51(1):1702052. doi: 10.1183/13993003.02052-2017. Print 2018 Jan. PMID 29371383
- [Background] Aksamit T, De Soyza A, Bandel TJ, Criollo M, Elborn JS, Operschall E, Polverino E, Roth K, Winthrop KL, Wilson R. RESPIRE 2: a phase III placebo-controlled randomised trial of ciprofloxacin dry powder for inhalation in non-cystic fibrosis bronchiectasis. Eur Respir J. 2018 Jan 25;51(1):1702053. doi: 10.1183/13993003.02053-2017. Print 2018 Jan. PMID 29371384
- [Background] Araujo D, Shteinberg M, Aliberti S, Goeminne PC, Hill AT, Fardon TC, Obradovic D, Stone G, Trautmann M, Davis A, Dimakou K, Polverino E, De Soyza A, McDonnell MJ, Chalmers JD. The independent contribution of Pseudomonas aeruginosa infection to long-term clinical outcomes in bronchiectasis. Eur Respir J. 2018 Jan 31;51(2):1701953. doi: 10.1183/13993003.01953-2017. Print 2018 Feb. PMID 29386336
- [Background] Wang H, Ji XB, Mao B, Li CW, Lu HW, Xu JF. Pseudomonas aeruginosa isolation in patients with non-cystic fibrosis bronchiectasis: a retrospective study. BMJ Open. 2018 Mar 14;8(3):e014613. doi: 10.1136/bmjopen-2016-014613. PMID 29540404
- [Background] Martinez-Garcia MA, Olveira C, Maiz L, Giron RM feminine, Prados C, de la Rosa D, Blanco M, Agusti A. Bronchiectasis: A Complex, Heterogeneous Disease. Arch Bronconeumol (Engl Ed). 2019 Aug;55(8):427-433. doi: 10.1016/j.arbres.2019.02.024. Epub 2019 Apr 18. English, Spanish. PMID 31005356
- [Background] O'Neill K, Einarsson GG, Rowan S, McIlreavey L, Lee AJ, Lawson J, Lynch T, Horsley A, Bradley JM, Elborn JS, Tunney MM. Composition of airway bacterial community correlates with chest HRCT in adults with bronchiectasis. Respirology. 2020 Jan;25(1):64-70. doi: 10.1111/resp.13653. Epub 2019 Jul 30. PMID 31364220
- [Background] Vermeersch K, Gabrovska M, Aumann J, Demedts IK, Corhay JL, Marchand E, Slabbynck H, Haenebalcke C, Haerens M, Hanon S, Jordens P, Peche R, Fremault A, Lauwerier T, Delporte A, Vandenberk B, Willems R, Everaerts S, Belmans A, Bogaerts K, Verleden GM, Troosters T, Ninane V, Brusselle GG, Janssens W. Azithromycin during Acute Chronic Obstructive Pulmonary Disease Exacerbations Requiring Hospitalization (BACE). A Multicenter, Randomized, Double-Blind, Placebo-controlled Trial. Am J Respir Crit Care Med. 2019 Oct 1;200(7):857-868. doi: 10.1164/rccm.201901-0094OC. PMID 31046405
- [Background] Serisier DJ, Martin ML, McGuckin MA, Lourie R, Chen AC, Brain B, Biga S, Schlebusch S, Dash P, Bowler SD. Effect of long-term, low-dose erythromycin on pulmonary exacerbations among patients with non-cystic fibrosis bronchiectasis: the BLESS randomized controlled trial. JAMA. 2013 Mar 27;309(12):1260-7. doi: 10.1001/jama.2013.2290. PMID 23532242
- [Background] Wang D, Fu W, Dai J. Meta-analysis of macrolide maintenance therapy for prevention of disease exacerbations in patients with noncystic fibrosis bronchiectasis. Medicine (Baltimore). 2019 Apr;98(17):e15285. doi: 10.1097/MD.0000000000015285. PMID 31027086
- [Background] Hodge S, Reynolds PN. Low-dose azithromycin improves phagocytosis of bacteria by both alveolar and monocyte-derived macrophages in chronic obstructive pulmonary disease subjects. Respirology. 2012 Jul;17(5):802-7. doi: 10.1111/j.1440-1843.2012.02135.x. PMID 22288725
- [Background] Wong C, Jayaram L, Karalus N, Eaton T, Tong C, Hockey H, Milne D, Fergusson W, Tuffery C, Sexton P, Storey L, Ashton T. Azithromycin for prevention of exacerbations in non-cystic fibrosis bronchiectasis (EMBRACE): a randomised, double-blind, placebo-controlled trial. Lancet. 2012 Aug 18;380(9842):660-7. doi: 10.1016/S0140-6736(12)60953-2. PMID 22901887
- [Background] Hill AT, Sullivan AL, Chalmers JD, De Soyza A, Elborn JS, Floto RA, Grillo L, Gruffydd-Jones K, Harvey A, Haworth CS, Hiscocks E, Hurst JR, Johnson C, Kelleher WP, Bedi P, Payne K, Saleh H, Screaton NJ, Smith M, Tunney M, Whitters D, Wilson R, Loebinger MR. British Thoracic Society guideline for bronchiectasis in adults. BMJ Open Respir Res. 2018 Dec 28;5(1):e000348. doi: 10.1136/bmjresp-2018-000348. eCollection 2018. PMID 30687502
- [Background] Polverino E, Goeminne PC, McDonnell MJ, Aliberti S, Marshall SE, Loebinger MR, Murris M, Canton R, Torres A, Dimakou K, De Soyza A, Hill AT, Haworth CS, Vendrell M, Ringshausen FC, Subotic D, Wilson R, Vilaro J, Stallberg B, Welte T, Rohde G, Blasi F, Elborn S, Almagro M, Timothy A, Ruddy T, Tonia T, Rigau D, Chalmers JD. European Respiratory Society guidelines for the management of adult bronchiectasis. Eur Respir J. 2017 Sep 9;50(3):1700629. doi: 10.1183/13993003.00629-2017. Print 2017 Sep. PMID 28889110